CLINICAL TRIAL: NCT04573101
Title: An EEG-based Exploration of the Variables Affecting Cortical Responses to Arabic Music Scales for a Personalised and Effective Music Therapy in the Middle East: a Clinical Study
Brief Title: EEG Responses to Arabic Music Scales
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Cornell Medical College in Qatar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 19-00013
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Healthy
Keywords: Music; Emotions; Ethnicity; Culture; Music Preference

STUDY DESIGN:
Intervention Model Description: Each participants is exposed to 24 different audio recordings and asked to select emotion that best describes feeling after each auditory stimulus. The 24 audio stimuli are distributed in a random manner by computer. In addition, emotional assessment is performed before and after the session. This is a total of 26 arms.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (26):
- Before intervention (No Intervention): Participants answer questionnaire before any stimulus is given.
- After intervention (No Intervention): Participants answer questionnaire after the series of stimulus is given.
- N1 (Ney - Improvisation- Saba Re) (Experimental): Improvisation with Ney, on Saba maqam on Re.
  Interventions: Other: Music listening / EEG recording
- O1 (Oud - Improvisation- Saba Re) (Experimental): Improvisation with Oud, on Saba maqam on Re.
  Interventions: Other: Music listening / EEG recording
- Q1(Qanun - Improvisation- Saba Re) (Experimental): Improvisation with Qanun, on Saba maqam on Re.
  Interventions: Other: Music listening / EEG recording
- N2 (Ney - Improvisation- Saba Sol) (Experimental): Improvisation with Ney, on Saba maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- O2 (Oud - Improvisation- Saba Sol) (Experimental): Improvisation with Oud, on Saba maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- Q2 (Qanun - Improvisation- Saba Sol) (Experimental): Improvisation with Qanun, on Saba maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- N3 (Ney - Improvisation- Kurd Re) (Experimental): Improvisation with Ney, on Kurd maqam on Re.
  Interventions: Other: Music listening / EEG recording
- O3 (Oud - Improvisation- Kurd Re) (Experimental): Improvisation with Oud, on Kurd maqam on Re.
  Interventions: Other: Music listening / EEG recording
- Q3 (Qanun - Improvisation- Kurd Re) (Experimental): Improvisation with Qanun, on Kurd maqam on Re.
  Interventions: Other: Music listening / EEG recording
- N4 (Ney - Improvisation- Kurd Sol) (Experimental): Improvisation with Ney, on Kurd maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- O4 (Oud - Improvisation- Kurd Sol) (Experimental): Improvisation with Oud, on Kurd maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- Q4 (Qanun - Improvisation- Kurd Sol) (Experimental): Improvisation with Qanun, on Kurd maqam on Sol.
  Interventions: Other: Music listening / EEG recording
- N5 (Ney - Known music- Kurd Re) (Experimental): Known music with Ney, on Kurd maqam on Re. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- O5 (Oud - Known music- Kurd Re) (Experimental): Known music with Oud, on Kurd maqam on Re. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- Q5 (Qanun - Known music- Kurd Re) (Experimental): Known music with Qanun, on Kurd maqam on Re. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- N6 (Ney - Known music- Kurd Sol) (Experimental): Known music with Ney, on Kurd maqam on Sol. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- O6 (Oud - Known music- Kurd Sol) (Experimental): Known music with Oud, on Kurd maqam on Sol. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- Q6 (Qanun - Known music- Kurd Sol) (Experimental): Known music with Qanun, on Kurd maqam on Sol. (El Rabii)
  Interventions: Other: Music listening / EEG recording
- N7 (Ney - Known music- Saba Re) (Experimental): Known music with Ney, on Saba maqam on Re. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording
- O7 (Oud - Known music- Saba Re) (Experimental): Known music with Oud, on Saba maqam on Re. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording
- Q7 (Qanun - Known music- Saba Re) (Experimental): Known music with Qanun, on Saba maqam on Re. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording
- N8 (Ney - Known music- Saba Sol) (Experimental): Known music with Ney, on Saba maqam on Sol. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording
- O8 (Oud - Known music- Saba Sol) (Experimental): Known music with Oud, on Saba maqam on Sol. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording
- Q8 (Qanun - Known music- Saba Sol) (Experimental): Known music with Qanun, on Saba maqam on Sol. (Howa Sahih)
  Interventions: Other: Music listening / EEG recording

INTERVENTIONS:
Other: Music listening / EEG recording — Participants listen to 24 different audio clips of 1 min long each, and select emotion in between. EEG is recorded while participants are listening. Participants select the emotion that best describes their feeling from Table 1 of the PANAS-X. https://www2.psychology.uiowa.edu/faculty/clark/panas-x.pdf
  Arms: N1 (Ney - Improvisation- Saba Re); N2 (Ney - Improvisation- Saba Sol); N3 (Ney - Improvisation- Kurd Re); N4 (Ney - Improvisation- Kurd Sol); N5 (Ney - Known music- Kurd Re); N6 (Ney - Known music- Kurd Sol); N7 (Ney - Known music- Saba Re); N8 (Ney - Known music- Saba Sol); O1 (Oud - Improvisation- Saba Re); O2 (Oud - Improvisation- Saba Sol); O3 (Oud - Improvisation- Kurd Re); O4 (Oud - Improvisation- Kurd Sol); O5 (Oud - Known music- Kurd Re); O6 (Oud - Known music- Kurd Sol); O7 (Oud - Known music- Saba Re); O8 (Oud - Known music- Saba Sol); Q1(Qanun - Improvisation- Saba Re); Q2 (Qanun - Improvisation- Saba Sol); Q3 (Qanun - Improvisation- Kurd Re); Q4 (Qanun - Improvisation- Kurd Sol); Q5 (Qanun - Known music- Kurd Re); Q6 (Qanun - Known music- Kurd Sol); Q7 (Qanun - Known music- Saba Re); Q8 (Qanun - Known music- Saba Sol)

SUMMARY:
Recent studies showed that various factors can contribute to the efficiency of a music therapy such as the type of music used, the type of instrument, the ethnicity, musical preference of the subjects and many others. Investigators noticed that most of studies and clinical trials, while acknowledging the importance of ethnicity and musical preferences, use the Western Music type in their investigations and practice. While in the Middle East, Music Therapy played a tremendous role in the 10th century since the "scales theory" of the famous Scientists El Farabi and Avicenna, very little countries of the Middle East are investing in scientific studies using Arabic Music as a therapeutic tool. This study will be an electroencephalogram (EEG)-based investigation on correlations of multiple factors that can influence the cortical responses of the subject to the music and self-reported state of emotion and anxiety.

DETAILED DESCRIPTION:
This is the first clinical study involving Music in Qatar and the Gulf region, and the first study to explore Arab Music Scales using a combination of EEG and self-reported assessements.

Using EEG, investigators will analyze the full brain activity of brainwaves produced by up to 100 subjects in response to the audio musical stimuli. 24 different audio recordings have been designed to investigate on different acoustic cues:

* with versus without quartertones
* known music versus improvisation
* Maqam Saba (sad) versus maqam Kurd (happy)
* 3 different Middle Eastern instruments: Ney, Oud and Qanun
* Two pitches: from Re or from Sol

The presentation of the audio stimuli clips will be randomized by the SuperLab5 software and EEG brainwaves will be recorded using the Power Lab (AD instrument). Between every audio clip, recording will be paused to ask the subjects to self-report on their emotional and anxiety states using a self-evaluation questionnaire. Subjects will be randomly assigned to morning of afternoon sessions of recording.

Using bioinformatic tools, investigators will perform a correlation study between EEG results, emotional self-report from the PANAS-X questionnaire, as well as answers to another questionnaire asking for their age, gender, ethnicity, right or left handedness, musical preferences, and if the subject plays an instrument.

The outcomes will have direct applications on the development of personalized Music Therapy in the region for treatment and management of mental health conditions, neurodegenerative diseases and other conditions that are of high prevalence in the region.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 years old to or above (might include pregnant women)
2. Living in Qatar
3. Understand either English or arabic

Exclusion Criteria:

1. Individuals not meeting the inclusion criteria
2. Individuals with auditory impairments
3. Individuals with any known neurological condition (including epilepsy, Alzheimer, Parkinson, Autism etc)
4. Individuals not able to come to the site (WCMQ).
5. Adults not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

PRIMARY OUTCOMES:
Quantification of brain waves | During the intervention (an average of 30 minutes)
  Relative power of each of the brainwaves (alpha, beta, gamma, theta, delta).
Quantification of selected emotions | immediately before each intervention
  Count of every emotion (selected by participant from the provided Table).
Quantification of selected emotions | immediately after each intervention
  Count of every emotion (selected by participant from the provided Table)

CONTACTS AND LOCATIONS:
Overall Officials: GHIZLANE BENDRISS, PhD, Principal Investigator — Weill Cornell Medicine Qatar
Locations (1):
- Ghizlane Bendriss, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Yes
Individual participants data that underlie the results reported will be available after deidentification beginning 3 months after publication and ending 3 years after publication. The study protocol and statistical analysis plan will also be available beginning 3 months after publication and ending 3 years after publication. Anyone who wishes to access the individual data, to achieve aims in the approved proposal, will be eligible to gain access to data by submitting a proposal to ghb2002@qatar-med.cornell.edu and data will be available at this link: https://drive.google.com/drive/folders/1OVjWK7RNTs18c4OIDQErzGjbhmUC98qi?usp=sharing
Supporting Information: Study Protocol, SAP
Time Frame: 3 month after publication and ending 3 years after publication.
Access Criteria: Send proposal to ghb2002@qatar-med.cornell.edu